CLINICAL TRIAL: NCT04004481
Title: Metabolites of Tramadol in the Postoperative Surgical Patients Admitted in the ICU
Brief Title: Metabolites of Tramadol in the Postoperative Surgical Patients
Acronym: METRAS
Status: Completed | Type: Observational
Sponsor: Osijek University Hospital (Other)
Collaborators: Josip Juraj Strossmayer University of Osijek (Other)
Responsible Party: Sponsor
Other Study IDs: OsijekUH
Record Dates: First submitted 2019-06-25; First posted 2019-07-02 (Actual); Results first posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Abdominal Surgery; Respiratory Failure; Renal Failure; Liver Dysfunction; Multiorgan Failure
Keywords: Tramadol; CYP2D6 polymorphism; analgesia; intensive care; organ failure
MeSH Terms: conditions — Respiratory Insufficiency; Renal Insufficiency; Liver Diseases; Multiple Organ Failure; Agnosia | interventions — Morphine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — CYP2D6 polymorphism will be done from DNA isolated from white cells.

GROUPS / COHORTS (1):
- Adult patients undergoing major open abdominal surgery: Observational study. In the patients undergoing major open abdominal surgery for cancer tramadol will be used for postoperative analgesia. In the postoperative period parent compound and metabolites of tramadol will be measured. Postoperative analgesia and adverse effects will be registered and compared between CYP2D6 phenotypes observed.
  Interventions: Drug: Postoperative analgesia using tramadol

INTERVENTIONS:
Drug: Postoperative analgesia using tramadol — Tramadol 100 mg will be given to the patients in the postoperative period.
  Other Names: Morphine for rescue analgesia

SUMMARY:
Tramadol is opioid analgesic widely used to treat moderate to severe pain. It is metabolized by cytochrome CYP2D6 into two major metabolites: pharmacologically active metabolite O-desmethyltramadol (M1) and inactive N-desmethyltramadol (M2), respectively. Tramadol kinetics in a population of patients undergoing major abdominal surgical procedures, and in patients with a greater or lesser degree of organic failure, is still not well researched. The investigators will measure plasma concentrations of tramadol and its metabolites after usual tramadol doses in ICU patients after major abdominal surgery. Also analgesic affect and side effect of tramadol will be recorded.

DETAILED DESCRIPTION:
The blood samples for the CYP2D6 gene polymorphism analysis will be taken from all patients included in the study. The patients will be categorized as slow (PM), normal (NM) or ultra-fast metabolizers (UM) of tramadol using analysis of the CYP2D6 phenotype. Standard laboratory findings including red blood cells, urea, creatinine, and cholinesterase will be done before surgery.

The patients will receive 500 mg of tramadol intravenously divided into 5 doses during the first 24 postoperative hours in the ICU. The plasma concentrations of tramadol, O-desmethyltramadol and N-desmethyltramadol will be measured 1, 2 and 4 hours after the first dose, and immediately before the 2nd, 3rd and 5th dose. There will therefore be 6 measurements of tramadol and its metabolites.

The analgesic effect of tramadol will be measured in awake patients with Numeric Rating Scale - NRS (0 - without pain, 10 - strong pain) 30 minutes before and 30 minutes after tramadol administration. The NRS value of 3 or less will be considered as adequate analgesia. In case of inadequate analgesia rescue analgesic (morphine) will be used according to the local protocol.

In unconscious patients the analgesic effect of tramadol will be tested by Critical Care Pain Observation Tool (CPOT). The CPOT value of less than 2 will be considered as adequate analgesia. In case of inadequate analgesia rescue analgesic (morphine) will be used according to the local protocol. During the first 24 hours side effect of tramadol, such as nausea, vomiting and new respiratory depression will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients after major abdominal surgery will be observed.
* surgical interventions requiring a laparotomy and involving resection of the organs of the digestive system
* postoperative ICU admission.

Exclusion Criteria:

* allergic reaction to tramadol
* patients under 18 years old
* patient over 90 years old
* BMI <18 and >35
* laparoscopic surgery
* chronic therapy with tramadol, cimetidine, paroxetine, pimozide, metoclopramide, amiodarone, olanzapine, chlorpromazine, fluphenazine, haloperidol, thioridazine, risperidone and clozapine

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients undergoing major open abdominal cancer surgery in Osijek University Hospital who are admitted in the ICU after surgery, age between 18 and 90 years, BMI >18 and <35, who signed the informed consent will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-03-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nenad Neskovic, MD, Principal Investigator — Osijek University Hospital
Locations (1):
- University Hospital Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yang Y, Botton MR, Scott ER, Scott SA. Sequencing the CYP2D6 gene: from variant allele discovery to clinical pharmacogenetic testing. Pharmacogenomics. 2017 May;18(7):673-685. doi: 10.2217/pgs-2017-0033. Epub 2017 May 4. PMID 28470112
- [Background] Qiao W, Yang Y, Sebra R, Mendiratta G, Gaedigk A, Desnick RJ, Scott SA. Long-Read Single Molecule Real-Time Full Gene Sequencing of Cytochrome P450-2D6. Hum Mutat. 2016 Mar;37(3):315-23. doi: 10.1002/humu.22936. Epub 2015 Dec 18. PMID 26602992
- [Background] Grond S, Sablotzki A. Clinical pharmacology of tramadol. Clin Pharmacokinet. 2004;43(13):879-923. doi: 10.2165/00003088-200443130-00004. PMID 15509185
- [Background] de Moraes NV, Lauretti GR, Coelho EB, Godoy AL, Neves DV, Lanchote VL. Impact of fraction unbound, CYP3A, and CYP2D6 in vivo activities, and other potential covariates to the clearance of tramadol enantiomers in patients with neuropathic pain. Fundam Clin Pharmacol. 2016 Apr;30(2):153-61. doi: 10.1111/fcp.12168. Epub 2015 Dec 11. PMID 26947771
- [Background] Xu J, Zhang XC, Lv XQ, Xu YY, Wang GX, Jiang B, Cai L, Cai XJ. Effect of the cytochrome P450 2D6*10 genotype on the pharmacokinetics of tramadol in post-operative patients. Pharmazie. 2014 Feb;69(2):138-41. PMID 24640604
- [Background] Stamer UM, Musshoff F, Kobilay M, Madea B, Hoeft A, Stuber F. Concentrations of tramadol and O-desmethyltramadol enantiomers in different CYP2D6 genotypes. Clin Pharmacol Ther. 2007 Jul;82(1):41-7. doi: 10.1038/sj.clpt.6100152. Epub 2007 Mar 14. PMID 17361124
- [Background] Candiotti KA, Birnbach DJ, Lubarsky DA, Nhuch F, Kamat A, Koch WH, Nikoloff M, Wu L, Andrews D. The impact of pharmacogenomics on postoperative nausea and vomiting: do CYP2D6 allele copy number and polymorphisms affect the success or failure of ondansetron prophylaxis? Anesthesiology. 2005 Mar;102(3):543-9. doi: 10.1097/00000542-200503000-00011. PMID 15731591
- [Background] Bosilkovska M, Walder B, Besson M, Daali Y, Desmeules J. Analgesics in patients with hepatic impairment: pharmacology and clinical implications. Drugs. 2012 Aug 20;72(12):1645-69. doi: 10.2165/11635500-000000000-00000. PMID 22867045
- [Background] Rijkenberg S, Stilma W, Bosman RJ, van der Meer NJ, van der Voort PHJ. Pain Measurement in Mechanically Ventilated Patients After Cardiac Surgery: Comparison of the Behavioral Pain Scale (BPS) and the Critical-Care Pain Observation Tool (CPOT). J Cardiothorac Vasc Anesth. 2017 Aug;31(4):1227-1234. doi: 10.1053/j.jvca.2017.03.013. Epub 2017 Mar 15. PMID 28800982
- [Background] Severgnini P, Pelosi P, Contino E, Serafinelli E, Novario R, Chiaranda M. Accuracy of Critical Care Pain Observation Tool and Behavioral Pain Scale to assess pain in critically ill conscious and unconscious patients: prospective, observational study. J Intensive Care. 2016 Nov 7;4:68. doi: 10.1186/s40560-016-0192-x. eCollection 2016. PMID 27833752
- [Derived] Neskovic N, Mandic D, Marczi S, Skiljic S, Kristek G, Vinkovic H, Mraovic B, Debeljak Z, Kvolik S. Different Pharmacokinetics of Tramadol, O-Demethyltramadol and N-Demethyltramadol in Postoperative Surgical Patients From Those Observed in Medical Patients. Front Pharmacol. 2021 Apr 15;12:656748. doi: 10.3389/fphar.2021.656748. eCollection 2021. PMID 33935773

RESULTS

PARTICIPANT FLOW:
Groups:
- Adult Patients Undergoing Major Open Abdominal Surgery: Observational study. In the patients undergoing major open abdominal surgery tramadol will be used for postoperative analgesia. In the postoperative period parent compound and metabolites of tramadol will be measured. Postoperative analgesia and adverse effects will be registered and compared between CYP2D6 phenotypes observed and in regards to systemic inflammation and preoperative cholinesterase activity.
  Postoperative analgesia using tramadol: Tramadol 100 mg will be given to the patients in the postoperative period.
Period: Overall Study
Arm/Group | Adult Patients Undergoing Major Open Abdominal Surgery
Started | 50
Completed | 47
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Adult Patients Undergoing Major Open Abdominal Surgery
Number analyzed (Participants) | 47
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 67 [59 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 47
  More than one race | 0
  Unknown or Not Reported | 0
Body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 26.1 [22.9 to 28.7]
ASA status [Count of Participants; unit: Participants] — ASA I: A normal healthy patient; ASA II: A patient with mild systemic disease; ASA III: A patient with severe systemic disease; ASA IV: A patient with severe systemic disease that is a constant threat to life; ASA V: A moribund patient who is not expected to survive without the operation.
  Participants
    ASA II | 11
    ASA III | 27
    ASA IV | 8
    ASA V | 1
CYP2D6 polymorphism [Count of Participants; unit: Participants]
  *1/*4 | 16
  *1/*1 | 22
  *1/*4xN | 3
  *4/*4 | 2
  *1/*3 | 2
  *1/*1xN | 1
Metabolic phenotype [Count of Participants; unit: Participants] — Metabolic phenotype was determined according to the CYP2D6 diplotype polymorphism.
  Participants
    Poor | 2
    Intermediate | 22
    Extensive | 22
    Ultrafast | 1

OUTCOME MEASURES:

1. Primary Outcome: Serum Concentration of Tramadol and Tramadol Metabolites With Respect to Metabolic Phenotype
Description: The plasma concentrations of tramadol, O-desmethyltramadol (ODT) and N-desmethyltramadol (NDT) will be measured 1, 2 and 4 hours after the first dose of 100 mg tramadol i.v., and immediately before the 2nd, 3rd and 5th dose. There will therefore be 6 measurements of tramadol and its metabolites.
Time Frame: 1, 2, and 4 hours after first dose and immediately before 2nd, 3rd, and 5th dose, up to 24 hours
Measure: Median (Inter-Quartile Range); unit: mcg/L
Groups:
- Tramadol Concentration: Median of tramadol concentration in 6 measurements point in postoperative 24 hours
- ODT Concentration in Poor Metabolizers (PM): Median ODT concentration in 6 measurements point in postoperative 24 hours in PM
- ODT Concentration in Intermediate Metabolizers (IM): Median ODT concentration in 6 measurements point in postoperative 24 hours in IM
- ODT Concentration in Extensive Metabolizers (EM): Median ODT concentration in 6 measurements point in postoperative 24 hours in EM
- ODT Concentration in Ultrafast Metabolizers (UM): Median ODT concentration in 6 measurements point in postoperative 24 hours in UM
- NDT Concentration in Poor Metabolizers (PM): Median NDT concentration in 6 measurements point in postoperative 24 hours in PM
- NDT Concentration in Intermediate Metabolizers (IM): Median NDT concentration in 6 measurements point in postoperative 24 hours in IM
- NDT Concentration in Extensive Metabolizers (EM): Median NDT concentration in 6 measurements point in postoperative 24 hours in EM
- NDT Concentration in Ultrafast Metabolizers (UM): Median NDT concentration in 6 measurements point in postoperative 24 hours in UM
Arm/Group | Tramadol Concentration | ODT Concentration in Poor Metabolizers (PM) | ODT Concentration in Intermediate Metabolizers (IM) | ODT Concentration in Extensive Metabolizers (EM) | ODT Concentration in Ultrafast Metabolizers (UM) | NDT Concentration in Poor Metabolizers (PM) | NDT Concentration in Intermediate Metabolizers (IM) | NDT Concentration in Extensive Metabolizers (EM) | NDT Concentration in Ultrafast Metabolizers (UM)
Number analyzed (Participants) | 47 | 2 | 22 | 22 | 1 | 2 | 22 | 22 | 1
mcg/L
  1st measurement | 372.7 [250.6 to 535.7] | 7.05 [4.52 to 7.05] | 17.1 [6.3 to 38.1] | 40.9 [21.9 to 53.9] | 13.8 | 11.7 [7.6 to 11.7] | 4.5 [3.5 to 11.1] | 4.76 [3.5 to 19.1] | 3.5
  2nd measurement | 270.6 [201.6 to 447.9] | 7.6 [4.5 to 7.6] | 15.7 [7.3 to 39.6] | 46.7 [23.6 to 64.3] | 19.4 | 15.3 [9.2 to 15.3] | 6.1 [3.9 to 12.2] | 5.2 [3.5 to 22] | 3.5
  3rd measurement | 232.1 [153.5 to 369.8] | 10 [4.6 to 10] | 20.2 [12.5 to 40.4] | 46.4 [31 to 72.6] | 26 | 28.9 [12.3 to 28.9] | 9.1 [5.3 to 14.7] | 8.5 [3.6 to 22.9] | 3.5
  4th measurement | 181.2 [122.9 to 270.2] | 12.4 [5.2 to 12.4] | 19.1 [11.4 to 47.8] | 38.1 [30.3 to 74.5] | 25.1 | 31.2 [15.7 to 31.2] | 9.6 [5.1 to 20.7] | 9.7 [3.5 to 23.9] | 3.5
  5th measurement | 300.1 [191.8 to 417.6] | 19.1 [10.7 to 19.1] | 36.6 [21.2 to 71.4] | 75.1 [46.3 to 117.6] | 58.2 | 71.4 [43 to 71.4] | 20.2 [10.5 to 37.2] | 19 [7.4 to 45.6] | 9.8
  6th measurement | 408.5 [273.8 to 677.8] | 29.7 [23.9 to 29.7] | 51.7 [25.7 to 93.5] | 97.4 [52.6 to 139] | 61.9 | 180.5 [124.9 to 180.5] | 34.9 [18.5 to 69.9] | 34.4 [18.6 to 72.5] | 18.1

2. Secondary Outcome: Analgesic Effect of Tramadol Measured by Numeric Rating Scale (NRS)
Description: The analgesic effect of tramadol will be measured in awake patients with Numeric Rating Scale (NRS, 0 - without pain, 10 - the worst pain) 30 minutes before and 30 minutes after tramadol administration. The NRS value of 3 or less will be considered as adequate analgesia. In case of inadequate analgesia morphine will be used according to the local protocol.
Time Frame: Before each dose of tramadol and 30 minutes after tramadol dose, up to 24 hours
Population: Pain was assessed by the NRS scale in patients who were awake.
Measure: Median (Inter-Quartile Range); unit: score on scale
Groups:
- Median NRS Score Before Tramadol Administration: NRS score value in awake patients before tramadol administration in 5 measurement point
- Median NRS Score After Tramadol Administration: NRS score value in awake patients after tramadol administration in 5 measurement point
Arm/Group | Median NRS Score Before Tramadol Administration | Median NRS Score After Tramadol Administration
Number analyzed (Participants) | 45 | 44
score on scale
  1st pain assessment: number analyzed (Participants) | 9 | 13
  1st pain assessment | 7 [3 to 9] | 5 [3.5 to 6]
  2nd pain assessment: number analyzed (Participants) | 40 | 40
  2nd pain assessment | 5 [3 to 6.75] | 3 [1 to 4.75]
  3rd pain assessment: number analyzed (Participants) | 44 | 44
  3rd pain assessment | 3.5 [2.25 to 5] | 2 [1 to 3]
  4th pain assessment: number analyzed (Participants) | 44 | 43
  4th pain assessment | 4 [2 to 5] | 2 [1 to 4]
  5th pain assessment | 3 [2 to 5] | 2 [1 to 3]

3. Secondary Outcome: Analgesic Effect of Tramadol Measured by Critical Care Pain Observation Tool (CPOT)
Description: In unconsciousness patents, the analgesic effect of tramadol will be tested by Critical Care Pain Observation Tool (CPOT). Highest score on a scale is 8 (worst pain) and lowest is 0 (no pain). The CPOT value of less than 2 will be considered as adequate analgesia.
Time Frame: Pain was assessed before and 30 minutes after each tramadol dose, up to 24 hours.
Population: All unconscious patients had low CPOT values and were therefore not suitable for statistical analysis.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Median CPOT Score Before Tramadol Administration: CPOT score value in awake patients before tramadol administration in 5 measurement point
- Median CPOT Score After Tramadol Administration: CPOT score value in awake patients after tramadol administration in 5 measurement point
Arm/Group | Median CPOT Score Before Tramadol Administration | Median CPOT Score After Tramadol Administration
Number analyzed (Participants) | 39 | 34
score on a scale
  1st assessment point | 0 [0 to 0] | 0 [0 to 0]
  2nd assessment point: number analyzed (Participants) | 7 | 7
  2nd assessment point | 0 [0 to 0] | 0 [0 to 0]
  3rd assessment point: number analyzed (Participants) | 3 | 3
  3rd assessment point | 0 [0 to 0] | 0 [0 to 0]
  4th assessment point: number analyzed (Participants) | 39 | 4
  4th assessment point | 0 [0 to 0] | 0 [0 to 0]
  5th assessment point: number analyzed (Participants) | 39 | 2
  5th assessment point | 0 [0 to 0] | 0 [0 to 0]

4. Secondary Outcome: Number of Participants With Nausea and Vomiting After Tramadol
Description: Nausea and/or vomiting during treatment with tramadol in ICU will be recorded.
Time Frame: Nausea and vomiting was assessed during first 30 minutes after tramadol administration
Measure: Count of Participants; unit: Participants
Groups:
- PONV in EM; PONV in IM: We monitored the incidence of PONV with respect to metabolic phenotype.
Arm/Group | PONV in EM | PONV in IM
Number analyzed (Participants) | 22 | 22
Participants | 12 | 4

5. Secondary Outcome: Number of Patients With Respiratory Depression After Tramadol
Description: Respiratory depression after tramadol is considered to be any drop in saturation below 90% or drop in respiratory rate below 10/min.
Time Frame: Respiratory depression was observed up to 30 minutes after tramadol administration
Measure: Count of Participants; unit: Participants
Groups:
- Number of Patients With Postoperative Respiratory Depression: We examined the occurrence of tramadol-induced respiratory depression in the first 24 hours
Arm/Group | Number of Patients With Postoperative Respiratory Depression
Number analyzed (Participants) | 47
Participants | 0

6. Secondary Outcome: Length of ICU Stay
Description: Length of stay in ICU will be recorded and correlated with standard laboratory values and tramadol and metabolites concentration.
Time Frame: Up to 6 months
Measure: Median (Inter-Quartile Range); unit: days
Groups:
- Low Plasma Cholinesterase Activity: Preoperative plasma cholinesterase activity < 4244 U/L
- Normal Plasma Cholinesterase Activity: Preoperative plasma cholinesterase activity > 4244 U/L
Arm/Group | Low Plasma Cholinesterase Activity | Normal Plasma Cholinesterase Activity
Number analyzed (Participants) | 18 | 25
days | 1.5 [1 to 6] | 1 [1 to 1]

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Postoperative nausea and/or vomiting
Arm/Group | PONV in EM | PONV in IM
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 12/22 | 4/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PONV in EM (N=22) | PONV in IM (N=22)
PONV (Gastrointestinal disorders) | 12 (12) | 4 (4) — Postoperative nausea and/or vomiting

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT04004481/Prot_SAP_000.pdf